CLINICAL TRIAL: NCT00200408
Title: Assessment of Early Genetic Changes in Smokers
Status: Terminated | Type: Observational
Why Stopped: unable to obtain funding
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Richard V. Smith, MD, MOntefiore Medical Center
Other Study IDs: 04-01-008S
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Cancer of Head and Neck; Smoking
Keywords: cancer of head and neck; smoking
MeSH Terms: conditions — Head and Neck Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- smokers: college students who smoke
- non smokers: college students who don't smoke

SUMMARY:
This study will look at the genetic profile of cells taken from the oral cavity of healthy college students who smoke and who do not smoke cigarettes. This will be done using a small brush similar to that used in Pap tests for cervical cancer detection. Our aim is to determine if smoking causes early genetic changes in the DNA of these cells such as have been seen in the cells of cancerous tumors of the head and neck area and nearby healthy tissues. This will be correlated with data from subject questionnaires to assess tobacco use, and other behavior and demographic information.

DETAILED DESCRIPTION:
Our pilot study using cellular DNA (cDNA) microarrays to examine the buccal mucosa of smokers and non-smokers demonstrated that smokers could be separated from non-smokers based solely on the patterns of gene expression observed. We were able to identify 924 genes whose expression differs significantly between samples from smokers and non-smokers. Several genes were also shown to be either up or down regulated in our earlier research applying microarray analysis to head and neck cancer tumors. Many of these represent genes of possible interest as early molecular markers for head and neck carcinogenesis.

Aberrant methylation is an important event in the transcriptional silencing of candidate tumor suppressor genes in smoking associated malignancies. Furthermore, it is known that methylated CpG islands are the preferred binding site for benzo(a)pyrene diol epoxide and other carcinogens found in tobacco smoke. Binding of these compounds is known to cause DNA adducts and transversion mutations that are often observed in the aerodigestive tumors of smokers. New evidence suggests that specific DNA methylation events are directly linked to tobacco use. The ability to detect such molecular markers during screening of high risk groups would represent a significant advance in cancer screening and early detection. Our group has evaluated specimens to epigenetically profile CpG island hypermethylation in. head and neck squamous cell carcinoma ( HNSCC) tumor samples using a technique known as methylation specific restriction enzyme microarray analysis. This method will be used in this trial to detect alterations in global DNA methylation patterns in subjects who smoke compared to those who don't.

The objectives of this study are:

1. Test the hypothesis that there are specific genetic alterations, leading to gene expression profile changes, which will be detected in early smokers.
2. Test the hypothesis that early smokers will demonstrate alterations in global DNA methylation patterns compared to matched controls.
3. To analyze gene alterations and DNA methylation in college smokers over time through longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

College freshmen and sophomores

Smokers must be between the ages of 18 and 25

Smokers must have smoked regularly for at least 2 years and be currently smoking

Smokers must intend to stay in the New York area for at least 3 years.

Non-smokers must be non-users of marijuana -

Exclusion Criteria:

Current HIV/AIDS infection

Use of chewing tobacco

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy smokers and non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2004-03; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
alteration of gene expression profile | 2 yrs
  comparison of gene expression profiles between smokers and non-smokers

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Smith, MD, Study Chair — Montefiore Medical Center; Thomas Belbin, PhD, Principal Investigator — Albert Einstein College of Medicine; Nicholas Schlecht, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States